CLINICAL TRIAL: NCT02791230
Title: A PHASE 3 MULTICENTER, OPEN-LABEL STUDY TO EVALUATE THE SAFETY OF DAILY ORAL DOSING OF TAFAMIDIS MEGLUMINE (PF-06291826-83) 20 MG OR 80 MG [OR TAFAMIDIS (PF-06291826-00) 61 MG] IN SUBJECTS DIAGNOSED WITH TRANSTHYRETIN CARDIOMYOPATHY (ATTR-CM)
Brief Title: Long-term Safety of Tafamidis in Subjects With Transthyretin Cardiomyopathy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: B3461045; 2016-000868-42 (EudraCT Number)
Record Dates: First submitted 2016-06-01; First posted 2016-06-06 (Estimated); Results first posted 2025-02-03 (Actual); Last update posted 2025-02-03 (Actual); Status verified 2025-01

CONDITIONS: Transthyretin (TTR) Amyloid Cardiomyopathy
Keywords: amyloidosis; amyloid; transthyretin; TTR; ATTR-CM
MeSH Terms: conditions — Amyloid Neuropathies, Familial; Amyloidosis; Alzheimer Disease | interventions — tafamidis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Tafamidis (Experimental): Active treatment - 61 mg or if not available, tafamidis meglumine 80 mg
  Interventions: Drug: Tafamidis

INTERVENTIONS:
Drug: Tafamidis — Soft gel capsules administered once a day for 60 months

SUMMARY:
Open label study to evaluate tafamidis for the treatment of transthyretin cardiomyopathy

DETAILED DESCRIPTION:
Global Phase 3, open label long term extension safety study designed to obtain additional safety data for tafamidis meglumine 20 mg and 80 mg (or tafamidis 61 mg where available), and to continue to provide enrolled subjects with tafamidis for up to 60 months, or until subject has access to tafamidis for ATTR CM via prescription, whichever occurs first.

ELIGIBILITY:
Inclusion Criteria:

Cohort A: Completion of 30 months of study treatment on Pfizer Protocol B3461028

Cohort B: Patients in specific countries diagnosed with ATTR-CM who did not previously participate in Pfizer Study B3461028

Exclusion Criteria:

-Liver and/or heart transplant, or implanted cardiac mechanical assist device

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1733 (Actual)
Dates: Start 2016-06-13 (Actual); Primary Completion 2023-10-26 (Actual); Study Completion 2023-11-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (80):
- United States (41):
  - The Kirklin Clinic of UAB Hospital, Birmingham, Alabama
  - Cardiovascular Clinical Trials Unit (CCTU), Birmingham, Alabama
  - University Hospital, University of Alabama at Birmingham, Birmingham, Alabama
  - California Heart Center, Beverly Hills, California
  - Cedars-Sinai Medical Care Foundation, Beverly Hills, California
  - Altman Clinical Translational Research Institute, La Jolla, California
  - University of California, San Diego, La Jolla, California
  - Cedars-Sinai Medical Center, Los Angeles, California
  - University of California, San Diego Medical Center - Hillcrest, San Diego, California
  - Center Adv Lab Medicine, San Diego, California
  - UCSF Ambulatory Care Center, San Francisco, California
  - University of California, San Francisco, California
  - UCSF Cardiovascular Care and Prevention Center, San Francisco, California
  - Stanford University Hospital and Clinics, Stanford, California
  - Sylvester at Deerfield Beach, Deerfield Beach, Florida
  - University of Miami Hospital & Clinics/Sylvester Comprehensive Cancer Center, Miami, Florida
  - Northwestern Medical Group, Chicago, Illinois
  - Northwestern Memorial Hospital, Chicago, Illinois
  - Advocate Christ Medical Center, Oak Lawn, Illinois
  - University of Maryland, Baltimore, Baltimore, Maryland
  - Johns Hopkins University, Baltimore, Maryland
  - Boston Medical Center Investigational Pharmacy, Boston, Massachusetts
  - Boston Medical Center, Boston, Massachusetts
  - Boston University Medical Center, Boston, Massachusetts
  - Michigan Medicine,University of Michigan, Ann Arbor, Michigan
  - Mayo Clinic Hospital-Rochester, Rochester, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - Newark Beth Israel Medical Center, Newark, New Jersey
  - NYU Langone Health, New York, New York
  - Center for Advanced Cardiac Care, New York, New York
  - Columbia University Irving Medical Center, New York, New York
  - Duke University, Durham, North Carolina
  - Cleveland Clinic, Cleveland, Ohio
  - OHSU Center for Health and Healing, Portland, Oregon
  - OHSU Research Pharmacy Services, Portland, Oregon
  - Oregon Health & Science University, Portland, Oregon
  - Penn Presbyterian Medical Center, Philadelphia, Pennsylvania
  - Vanderbilt Univ. Med. Ctr, Nashville, Tennessee
  - Huntsman Cancer Hospital, Salt Lake City, Utah
  - University of Utah Hospitals & Clinics, Salt Lake City, Utah
  - University of Utah, Division of Cardiovascular Medicine, Salt Lake City, Utah
- Instituto Cardiovascular de Buenos Aires, Buenos Aires, Argentina
- Australia (3):
  - Westmead Hospital, Westmead, New South Wales
  - Princess Alexandra Hospital, Woolloongabba, Queensland
  - Eastern Health (Box Hill Hospital), Box Hill, Victoria
- UZ Leuven, Leuven, Belgium
- Hospital Universitário Clementino Fraga Filho (UFRJ), Rio de Janeiro, Rio de Janeiro, Brazil
- Canada (4):
  - University of Calgary/Foothills Medical Centre, Calgary, Alberta
  - Vancouver General Hospital, Vancouver, British Columbia
  - Toronto General Hospital, Toronto, Ontario
  - Montreal Heart Institute, Montreal, Quebec
- Czechia (3):
  - Fakultni nemocnice u sv. Anny v Brne, Brno
  - Vseobecna fakultni nemocnice v Praze, Prague
  - Institut klinicke a experimentalni mediciny, Prague
- France (7):
  - Hopital de La Timone, Marseille, CAN
  - CHU Henri Mondor, Créteil
  - Hôpital De La Timone, Marseille
  - Hopital Bichat, Paris
  - CHU de Rennes - Hopital Pontchaillou, Rennes
  - CHU de Rennes - Hôpital Pontchaillou, Rennes
  - CHU de Toulouse - Hôpital Rangueil, Toulouse
- Germany (2):
  - Medical University of Heidelberg, Heidelberg
  - Universitätsklinikum Münster, Münster
- Hong Kong (2):
  - Clinical Trial Pharmacy, Hong Kong
  - Queen Mary Hospital, Hong Kong
- Italy (3):
  - Azienda Ospedaliero-Universitaria Policlinico S. Orsola Malpighi, Bologna
  - Azienda Ospedaliero-Universitaria Careggi, Florence
  - Fondazione IRCCS Policlinico San Matteo, Pavia
- Japan (3):
  - Kurume University Hospital, Kurume-shi, Fukuoka
  - Kumamoto University Hospital, Kumamoto, Kumamoto
  - Shinshu University Hospital, Nagano
- University Medical Center Groningen, Groningen, Netherlands
- Spain (2):
  - Unidad de Insuficiencia Cardiaca Avanzada y Transplante Cardiaco, A Coruña, LA Coruna
  - Hospital Universitario Puerta de Hierro Majadahonda, Majadahonda, Madrid
- Sweden (2):
  - Skellefteå Lasarett, Skellefteå
  - Akademiska Sjukhuset, Uppsala
- Taiwan (3):
  - Investigational Drug Services, Taipei
  - National Taiwan University Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei
- Barts Health NHS Trust, St Bartholomew's Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- [Derived] Crespo-Leiro MG, Hanna M, Damy T, Delgado D, Ebede B, Marino V, Wang R, Maurer MS, Garcia-Pavia P, Drachman BM. Early Access to Tafamidis for Patients With Transthyretin Amyloid Cardiomyopathy. JACC Adv. 2025 Oct;4(10 Pt 2):102122. doi: 10.1016/j.jacadv.2025.102122. Epub 2025 Sep 10. PMID 40934814
- [Derived] Damy T, Wang R, Maurer MS, Gillmore JD, Fontana M. Long-term efficacy of tafamidis in patients with transthyretin amyloid cardiomyopathy by National Amyloidosis Centre stage. Eur J Heart Fail. 2025 Jun 9. doi: 10.1002/ejhf.3696. Online ahead of print. PMID 40488446
- [Derived] Drachman B, Damy T, Hanna M, Wang R, Angeli FS, Garcia-Pavia P. Long-term tafamidis efficacy in patients with transthyretin amyloid cardiomyopathy by baseline left ventricular ejection fraction. Eur J Heart Fail. 2024 Sep;26(9):2038-2046. doi: 10.1002/ejhf.3330. Epub 2024 Jun 26. PMID 38932583
- [Derived] Garcia-Pavia P, Sultan MB, Gundapaneni B, Sekijima Y, Perfetto F, Hanna M, Witteles R. Tafamidis Efficacy Among Octogenarian Patients in the Phase 3 ATTR-ACT and Ongoing Long-Term Extension Study. JACC Heart Fail. 2024 Jan;12(1):150-160. doi: 10.1016/j.jchf.2023.08.032. Epub 2023 Nov 8. PMID 37943223
- [Derived] Elliott P, Gundapaneni B, Sultan MB, Ines M, Garcia-Pavia P. Improved long-term survival with tafamidis treatment in patients with transthyretin amyloid cardiomyopathy and severe heart failure symptoms. Eur J Heart Fail. 2023 Nov;25(11):2060-2064. doi: 10.1002/ejhf.2974. Epub 2023 Jul 26. PMID 37434378
- [Derived] Elliott P, Drachman BM, Gottlieb SS, Hoffman JE, Hummel SL, Lenihan DJ, Ebede B, Gundapaneni B, Li B, Sultan MB, Shah SJ. Long-term survival in people with transthyretin amyloid cardiomyopathy who took tafamidis: A Plain Language Summary. Future Cardiol. 2023 Jan;19(1):7-17. doi: 10.2217/fca-2022-0096. Epub 2023 Jan 30. PMID 36715498
- [Derived] Elliott P, Drachman BM, Gottlieb SS, Hoffman JE, Hummel SL, Lenihan DJ, Ebede B, Gundapaneni B, Li B, Sultan MB, Shah SJ. Long-Term Survival With Tafamidis in Patients With Transthyretin Amyloid Cardiomyopathy. Circ Heart Fail. 2022 Jan;15(1):e008193. doi: 10.1161/CIRCHEARTFAILURE.120.008193. Epub 2021 Dec 20. PMID 34923848
- [Derived] Damy T, Garcia-Pavia P, Hanna M, Judge DP, Merlini G, Gundapaneni B, Patterson TA, Riley S, Schwartz JH, Sultan MB, Witteles R. Efficacy and safety of tafamidis doses in the Tafamidis in Transthyretin Cardiomyopathy Clinical Trial (ATTR-ACT) and long-term extension study. Eur J Heart Fail. 2021 Feb;23(2):277-285. doi: 10.1002/ejhf.2027. Epub 2020 Nov 12. PMID 33070419
- [Derived] Li B, Alvir J, Stewart M. Extrapolation of Survival Benefits in Patients with Transthyretin Amyloid Cardiomyopathy Receiving Tafamidis: Analysis of the Tafamidis in Transthyretin Cardiomyopathy Clinical Trial. Cardiol Ther. 2020 Dec;9(2):535-540. doi: 10.1007/s40119-020-00179-2. Epub 2020 Jun 10. PMID 32524297
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=B3461045

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study consisted of two cohorts: Cohort A and B. Cohort A: Participants diagnosed with transthyretin amyloid cardiomyopathy (ATTR-CM) who completed 30 months of participation in parent study [B3461028 (NCT01994889)] were enrolled in this current extension study (B3461045 [NCT02791230]). Cohort B: Participants diagnosed with ATTR-CM who did not participate in parent study B3461028 study were enrolled in this extension study.
Groups:
- Cohort A: Tafamidis (Parent and Extension Study): Eligible participants who received tafamidis in the parent study, after enrolment in the current extension study continued to receive tafamidis 61 milligrams (mg) or 80 mg (in regions where 61 mg tafamidis was unavailable), orally once daily along with standard of care for up to 60 months.
- Cohort A: Placebo (Parent Study)/Tafamidis (Extension Study): Eligible participants who received placebo in the parent study, after enrolment in the current extension study continued to receive tafamidis 61 mg or 80 mg (in regions where 61 mg tafamidis was unavailable), orally once daily along with standard of care for up to 60 months.
- Cohort B: Tafamidis (Only in Extension Study): Participants who did not participate in the parent study and received tafamidis at a dose of 61 mg (or 80 mg in regions where 61 mg tafamidis was unavailable), once daily along with standard of care for up to 60 months.
Period: Overall Study
Arm/Group | Cohort A: Tafamidis (Parent and Extension Study) | Cohort A: Placebo (Parent Study)/Tafamidis (Extension Study) | Cohort B: Tafamidis (Only in Extension Study)
Started | 170 | 82 | 1481
Treated | 170 | 82 | 1476
Completed | 84 | 31 | 988
Not Completed | 86 | 51 | 493
Not completed — Adverse Event | 10 | 9 | 66
Not completed — Death | 38 | 25 | 184
Not completed — Lack of Efficacy | 1 | 0 | 3
Not completed — Lost to Follow-up | 0 | 0 | 10
Not completed — Failure to Meet Randomization Criteria | 3 | 2 | 15
Not completed — Medication Error Without Associated Adverse Event | 0 | 1 | 1
Not completed — Study sites terminated by sponsor | 1 | 0 | 5
Not completed — Other | 9 | 1 | 28
Not completed — Protocol Violation | 0 | 0 | 4
Not completed — Withdrawal by Subject | 24 | 13 | 172
Not completed — Enrolled but not treated | 0 | 0 | 5

BASELINE CHARACTERISTICS:
Population: The safety analysis population consisted of all participants (Cohorts A and B) who were enrolled in this study and who had taken at least one dose of study treatment.
Groups:
- Cohort A: Tafamidis (Parent and Extension Study): Eligible participants who received tafamidis in the parent study, after enrolment in the current extension study continued to receive tafamidis 61 mg or 80 mg (in regions where 61 mg tafamidis was unavailable), orally once daily along with standard of care for up to 60 months.
- Total: Total of all reporting groups
Arm/Group | Cohort A: Tafamidis (Parent and Extension Study) | Cohort A: Placebo (Parent Study)/Tafamidis (Extension Study) | Cohort B: Tafamidis (Only in Extension Study) | Total
Number analyzed (Participants) | 170 | 82 | 1476 | 1728
Age, Continuous [Mean (Standard Deviation); unit: Years] | 76.73 (6.75) | 76.41 (6.47) | 76.51 (7.75) | 76.52 (7.60)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 8 | 165 | 186
  Male | 157 | 74 | 1311 | 1542
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 1 | 37 | 43
  Not Hispanic or Latino | 164 | 81 | 1433 | 1678
  Unknown or Not Reported | 1 | 0 | 6 | 7
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 9 | 5 | 66 | 80
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 15 | 5 | 139 | 159
  White | 144 | 72 | 1252 | 1468
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 2 | 0 | 19 | 21

OUTCOME MEASURES:

1. Primary Outcome: Time to All-Cause Mortality: Cohort A
Description: Time to all-cause mortality was calculated from first dose of randomized treatment in parent study (B3461028) to all-cause mortality events. All-cause mortality events included deaths, heart transplants and cardiac mechanical assist devices implantation treated as death. Treated participants from the parent study who discontinued prior to the start of this study were also included in this analysis as planned. Data from participants who dropped out for a liver-only transplantation were handled in the same manner as the data from all other censored participants. Censored participants were participants who completed study or discontinued from the study (including discontinued by sponsor or participants withdrew, or discontinued due to Adverse event (AE), or alive at the time of analysis. Kaplan Meier method was used for analysis. Therefore, this analysis was based on the pooled dose groups, as per the statistical analysis plan (SAP).
Time Frame: From first dose of randomized treatment in parent study (B3461028) up to 28 days post last dose of study treatment in current extension study (B3461045), [approximately up to 91 months]
Population: Combined mortality analysis (CMA) set included all participants in the Intent-To-Treat (ITT)-analysis set from study B3461028 (NCT01994889). Mortality analyses in study B3461045 for Cohort A participants included combined data from participants in study B3461028 (NCT01994889), including participants who died, discontinued in B3461028, or were not enrolled into B3461045 (i.e. ITT Analysis Set from B3461028 [NCT01994889]) with mortality data through participation in the B3461045 study.
Measure: Median (95% Confidence Interval); unit: Months
Groups:
- Cohort A: Tafamidis (Parent Study) and Tafamidis (Extension Study): Eligible participants who received tafamidis in the parent study, after enrolment in the current extension study continued to receive tafamidis 61 mg or 80 mg (in regions where 61 mg tafamidis was unavailable), orally once daily along with standard of care for up to 60 months.
- Cohort A: Placebo (Parent Study) and Tafamidis (Extension Study): Eligible participants who received placebo in the parent study, after enrolment in the current extension study continued to receive tafamidis 61 mg or 80 mg (in regions where 61 mg tafamidis was unavailable), orally once daily along with standard of care for up to 60 months.
Arm/Group | Cohort A: Tafamidis (Parent Study) and Tafamidis (Extension Study) | Cohort A: Placebo (Parent Study) and Tafamidis (Extension Study)
Number analyzed (Participants) | 264 | 177
Months | 58.7 [50.3 to 68.4] | 35.8 [29.7 to 41.1]
Statistical Analysis 1: Comparison: Cohort A: Tafamidis (Parent Study) and Tafamidis (Extension Study) vs Cohort A: Placebo (Parent Study) and Tafamidis (Extension Study); Test type: Superiority; p = 0.0001, Cox proportional hazards model; Hazard Ratio (HR) = 0.6202, 95% CI 2-sided [0.4865 to 0.7906] — Hazard ratio from a Cox proportional hazards model with treatment, Transthyretin (TTR) genotype (variant and wild-type) and New York Heart Association (NYHA) baseline classification (NYHA Classes I and II combined and NYHA Class III) in the model

2. Primary Outcome: Number of Participants With All-Cause Mortality Events: Cohort B
Description: All-cause mortality included all participants who had discontinue for transplantation (i.e. heart transplantation and combined heart and liver transplantation) or for implantation of a cardiac mechanical assist device, were handled in the same manner as death. Data from participants who dropped out for a liver-only transplantation were handled in the same manner as the data from all other censored participants. Censored participants were participants who completed study or discontinued from the study (including discontinued by sponsor or participants withdrew, or discontinued due to AE), or alive at the time of analysis. Kaplan Meier method was used for analysis.
Time Frame: B3461045: From first dose of treatment up to 28 days post last dose of study treatment (approximately up to 61 months)
Population: Safety analysis population consisted of all participants (Cohort B) who were enrolled in this study and who had taken at least 1 dose of study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort B: Tafamidis (Only in Extension Study)
Number analyzed (Participants) | 1476
Participants | 345

3. Primary Outcome: Number of Participants With Treatment-Emergent Adverse Events (AEs)
Description: An AE was any untoward medical occurrence in a participant who received investigational product or medical device; the event need not necessarily have a causal relationship with the treatment or usage. A treatment emergent AE was defined as an event that emerged during the treatment period that was absent before treatment or worsened during the treatment period relative to the pretreatment state. AEs included both SAEs and all Non-SAEs. A serious adverse event (SAE) was any untoward medical occurrence at any dose that: resulted in death; was life-threatening (immediate risk of death); required inpatient hospitalization or prolongation of existing hospitalization; resulted in persistent or significant disability/ incapacity; resulted in congenital anomaly/birth defect; considered an important medical event.
Time Frame: B3461045: From first dose of treatment up to 28 days post last dose of study treatment (approximately up to 61 months)
Population: Safety analysis population consisted of all participants (Cohorts A and B) who were enrolled in this study and taken at least 1 dose of study medication. Therefore, this analysis (Cohort A) was based on the pooled dose groups, as per the SAP.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A: Tafamidis (Parent and Extension Study) | Cohort A: Placebo (Parent Study)/Tafamidis (Extension Study) | Cohort B: Tafamidis (Only in Extension Study)
Number analyzed (Participants) | 170 | 82 | 1476
Participants | 168 | 79 | 1294

4. Other Pre Specified Outcome: Time to Cardiovascular-Related Mortality Events: Cohort A
Description: Time to cardiovascular-related mortality was calculated from first dose of randomized treatment in B3461028 . Participants who discontinued for transplantation (that is heart transplantation and combined heart and liver transplantation) or for implantation of cardiac mechanical assist device were treated as a death. Treated participants from the parent study who discontinued prior to the start of this study were also included in this analysis as planned. Kaplan-Meier method was used. Therefore, this analysis was based on the pooled dose groups, as per the SAP.
Time Frame: as for outcome 1
Population: CMA set included all participants in the ITT analysis set from study B3461028 (NCT01994889). Mortality analyses in study B3461045 for Cohort A participants were combined data from participants in study B3461028 (NCT01994889), including participants who died, discontinued in B3461028, or were not enrolled into B3461045 (i.e. ITT Analysis Set from B3461028 [NCT01994889]) with mortality data through participation in the B3461045 study.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Cohort A: Tafamidis (Parent Study) and Tafamidis (Extension Study) | Cohort A: Placebo (Parent Study) and Tafamidis (Extension Study)
Number analyzed (Participants) | 264 | 177
Months | 70.2 [63.4 to 88.8] | 40.8 [34.1 to 50.7]
Statistical Analysis 1: Comparison: Cohort A: Tafamidis (Parent Study) and Tafamidis (Extension Study) vs Cohort A: Placebo (Parent Study) and Tafamidis (Extension Study); Test type: Superiority; p = 0.0005, Cox Proportional Hazards model; Hazard ratio = 0.6133, 95% CI 2-sided [0.4666 to 0.8062] — Hazard ratio from a Cox proportional hazards model with treatment, TTR genotype (variant and wild-type) and NYHA baseline classification (NYHA Classes I and II combined and NYHA Class III) in the model

5. Other Pre Specified Outcome: Number of Participants With Cardiovascular Related Mortality Events: Cohort B
Description: Deaths adjudicated as cardiovascular-related and indeterminate were reported. Cardiovascular-related mortality events included deaths, heart transplants and cardiac mechanical assist devices implantation treated as death. Cardiovascular relatedness was based on clinical judgement.
Time Frame: B3461045: From first dose of treatment up to 28 days post last dose of study treatment (approximately up to 61 months)
Population: Safety analysis population included all participants who were enrolled in this study and taken at least 1 dose of study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort B: Tafamidis (Only in Extension Study)
Number analyzed (Participants) | 1476
Participants | 204

6. Other Pre Specified Outcome: Mean Annualized Rate of All Cause Hospitalizations
Description: Mean annual rate of all cause hospitalization was calculated for each participant as the participant's number of all cause hospitalizations divided by this participant's duration on study in years. Hospitalization was defined as any initial admission (even less than 24 hours) in a hospital or equivalent healthcare facility or any prolongation of an existing admission. Only all cause hospitalizations where the participant was admitted to a hospital during the current extension study were included in this analysis. Any hospitalizations prior to randomization date were not included.
Time Frame: B3461045: From first dose of treatment up to 28 days post last dose of study treatment (approximately up to 61 months)
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Hospitalization/year
Arm/Group | Cohort A: Tafamidis (Parent and Extension Study) | Cohort A: Placebo (Parent Study)/Tafamidis (Extension Study) | Cohort B: Tafamidis (Only in Extension Study)
Number analyzed (Participants) | 170 | 82 | 1476
Hospitalization/year | 1.67 (5.830) | 1.84 (2.275) | 0.96 (5.117)

7. Other Pre Specified Outcome: Mean Annualized Rate of Cardiovascular (CV)-Related Hospitalizations
Description: Mean annual rate of CV related hospitalization was calculated for each participant as the participant's number of CV related hospitalizations divided by this participant's duration on study in years. CV-related hospitalizations included hospitalizations due to heart failure, arrhythmia, myocardial infarction, stroke, and other cardiovascular-related events. Hospitalization was defined as any initial admission (even less than 24 hours) in a hospital or equivalent healthcare facility or any prolongation of an existing admission. Admission also included transfer within the hospital to an acute/intensive care unit (example: from the psychiatric wing to a medical floor, medical floor to a coronary care unit, or neurological floor to a tuberculosis unit).
Time Frame: B3461045: From first dose of treatment up to 28 days post last dose of study treatment (approximately up to 61 months)
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: CV related hospitalization/year
Arm/Group | Cohort A: Tafamidis (Parent and Extension Study) | Cohort A: Placebo (Parent Study)/Tafamidis (Extension Study) | Cohort B: Tafamidis (Only in Extension Study)
Number analyzed (Participants) | 170 | 82 | 1476
CV related hospitalization/year | 1.09 (5.409) | 1.14 (1.899) | 0.50 (1.567)

8. Other Pre Specified Outcome: Change From Baseline in Kansas City Cardiomyopathy Questionnaire (KCCQ) Clinical Summary Scores at Months 12, 30, 42, 60 and 90: Cohort A
Description: KCCQ: 23-item, self-administered questionnaire that assesses health status and health-related quality of life in participants with heart failure. KCCQ quantifies 8 domains: physical limitations, symptom stability, symptom frequency, symptom burden, total symptom (mean of symptom frequency and symptom burden), self-efficacy, quality of life and social limitations). Scores were generated for each domain and scaled from 0 (worst) to 100 (best possible status). KCCQ-clinical summary score was calculated as mean of the following domains- physical limitation and total symptoms and transformed to a single score which ranged from 0 (worst) -100 (best possible status), higher scores = better health status. Data for change from baseline was reported as least square (LS) mean.
Time Frame: B3461028: Baseline (Day 1, pre-dose), Months 12, 30; B3461045: Months 42, 60 and 90 (time points were relative to Day 1 from B3461028; 42, 60 and 90 Months were 12, 30 and 60 Months of B3461045)
Population: CMA set was analyzed. All participants reported under "Number of Participants Analyzed" contributed data to the table; however, may not have evaluable data for every row. "Number Analyzed" signifies number of participants evaluable at specified time points. Therefore, this analysis was based on the pooled dose groups, as per the SAP.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Cohort A: Tafamidis (Parent Study) and Tafamidis (Extension Study) | Cohort A: Placebo (Parent Study) and Tafamidis (Extension Study)
Number analyzed (Participants) | 264 | 177
Units on a scale
  Change at Month 12: number analyzed (Participants) | 221 | 145
  Change at Month 12 | -3.17 (1.016) | -10.2 (1.316)
  Change at Month 30: number analyzed (Participants) | 170 | 84
  Change at Month 30 | -7.41 (1.185) | -19.9 (1.999)
  Change at Month 42: number analyzed (Participants) | 143 | 54
  Change at Month 42 | -11.2 (1.483) | -25.4 (2.143)
  Change at Month 60: number analyzed (Participants) | 64 | 22
  Change at Month 60 | -11.8 (1.756) | -25.1 (3.287)
  Change at Month 90: number analyzed (Participants) | 9 | 2
  Change at Month 90 | -17.4 (2.758) | -56.9 (1.868)

9. Other Pre Specified Outcome: Change From Baseline in KCCQ Overall Score at Months 12, 30, 42, 60, 90: Cohort A
Description: KCCQ: 23-item, self-administered questionnaire that assesses health status and health-related quality of life in participants with heart failure. KCCQ quantifies 8 domains: physical limitations, symptom stability, symptom frequency, symptom burden, total symptom (mean of symptom frequency and symptom burden), self-efficacy, quality of life and social limitations). Scores were generated for each domain and scaled from 0 (worst) to 100 (best possible status). KCCQ-overall score was calculated as mean of the following domains- physical limitation, total symptoms (average of symptom frequency & symptom burden), quality of life, social limitation and transformed to a single score which ranged from 0 (worst) -100 (best possible status), higher scores = better health status. Data for change from baseline was reported as LS mean.
Time Frame: as for outcome 8
Population: as for outcome 8
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Cohort A: Tafamidis (Parent Study) and Tafamidis (Extension Study) | Cohort A: Placebo (Parent Study) and Tafamidis (Extension Study)
Number analyzed (Participants) | 264 | 177
Units on a scale
  Change at Month 12: number analyzed (Participants) | 221 | 145
  Change at Month 12 | -1.97 (1.131) | -9.69 (1.428)
  Change at Month 30: number analyzed (Participants) | 170 | 84
  Change at Month 30 | -6.07 (1.399) | -19.5 (1.908)
  Change at Month 42: number analyzed (Participants) | 143 | 54
  Change at Month 42 | -8.81 (1.470) | -24.0 (2.114)
  Change at Month 60: number analyzed (Participants) | 64 | 22
  Change at Month 60 | -8.56 (1.646) | -24.5 (3.020)
  Change at Month 90: number analyzed (Participants) | 9 | 2
  Change at Month 90 | -18.1 (2.617) | -52.6 (1.791)

10. Other Pre Specified Outcome: Change From Baseline in KCCQ Total Symptom Score at Months 12, 30, 42, 60 and 90: Cohort A
Description: KCCQ: 23-item, self-administered questionnaire that assesses health status and health-related quality of life in participants with heart failure. KCCQ quantifies 8 domains: physical limitations, symptom stability, symptom frequency, symptom burden, total symptom (mean of symptom frequency and symptom burden), self-efficacy, quality of life and social limitations). Scores were generated for each domain and scaled from 0 (worst) to 100 (best possible status). KCCQ Total Symptoms score was calculated as mean of the following domains- symptom frequency and symptom burden and transformed to a single score which ranged from 0 (worst) -100 (best possible status), higher scores = better health status. Data for change from baseline was reported as LS mean.
Time Frame: as for outcome 8
Population: as for outcome 8
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Cohort A: Tafamidis (Parent Study) and Tafamidis (Extension Study) | Cohort A: Placebo (Parent Study) and Tafamidis (Extension Study)
Number analyzed (Participants) | 264 | 177
Units on a scale
  Change at Month 12: number analyzed (Participants) | 221 | 145
  Change at Month 12 | -2.90 (1.182) | -10.3 (1.494)
  Change at Month 30: number analyzed (Participants) | 170 | 84
  Change at Month 30 | -5.92 (1.279) | -18.7 (2.276)
  Change at Month 42: number analyzed (Participants) | 143 | 54
  Change at Month 42 | -9.29 (1.699) | -22.5 (2.237)
  Change at Month 60: number analyzed (Participants) | 64 | 22
  Change at Month 60 | -8.94 (1.858) | -19.0 (3.693)
  Change at Month 90: number analyzed (Participants) | 9 | 2
  Change at Month 90 | -16.4 (2.654) | -56.0 (1.958)

11. Other Pre Specified Outcome: Change From Baseline in KCCQ Clinical Summary Scores at Months 12, 30 and 54: Cohort B
Description: KCCQ: 23-item, self-administered questionnaire that assesses health status and health-related quality of life in participants with heart failure. KCCQ quantifies 8 domains: physical limitations, symptom stability, symptom frequency, symptom burden, total symptom (mean of symptom frequency and symptom burden), self-efficacy, quality of life and social limitations). Scores were generated for each domain and scaled from 0 (worst) to 100 (best possible status). KCCQ-clinical summary score was calculated as mean of the following domains- physical limitation and total symptoms and transformed to a single score which ranged from 0 (worst) -100 (best possible status), higher scores = better health status. Data for change from baseline was reported as mean.
Time Frame: B3461045: Baseline (Day 1, pre-dose), Months 12, 30 and 54
Population: Safety analysis population included all participants (Cohort B) who were enrolled in this study and taken at least 1 dose of study medication. All participants reported under "Number of Participants Analyzed" contributed data to the table; however, may not have evaluable data for every row. Here, "Number Analyzed" signifies number of participants evaluable at specified time points.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Cohort B: Tafamidis (Only in Extension Study)
Number analyzed (Participants) | 830
Units on a scale
  Change at Month 12 | -0.242 (17.7032)
  Change at Month 30: number analyzed (Participants) | 237
  Change at Month 30 | -3.086 (20.4276)
  Change at Month 54: number analyzed (Participants) | 42
  Change at Month 54 | -3.988 (18.7931)

12. Other Pre Specified Outcome: Change From Baseline in KCCQ Overall Score at Months 12, 30 and 54: Cohort B
Description: KCCQ: 23-item, self-administered questionnaire that assesses health status and health-related quality of life in participants with heart failure. KCCQ quantifies 8 domains: physical limitations, symptom stability, symptom frequency, symptom burden, total symptom (mean of symptom frequency and symptom burden), self-efficacy, quality of life and social limitations). Scores were generated for each domain and scaled from 0 (worst) to 100 (best possible status). KCCQ-overall score was calculated as mean of the following domains- physical limitation, total symptoms (average of symptom frequency & symptom burden), quality of life, social limitation and transformed to a single score which ranged from 0 (worst) -100 (best possible status), higher scores = better health status. Data for change from baseline was reported as mean.
Time Frame: B3461045: Baseline (Day 1, pre-dose), Months 12, 30 and 54
Population: Safety analysis population included all participants (Cohort B) who were enrolled in this study and taken at least 1 dose of study medication. All participants reported under "Number of Participants Analyzed" contributed data to the table; however, may not have evaluable data for every row. "Number Analyzed" signifies number of participants evaluable at specified time points.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Cohort B: Tafamidis (Only in Extension Study)
Number analyzed (Participants) | 830
Units on a scale
  Change at Month 12 | 0.443 (18.2575)
  Change at Month 30: number analyzed (Participants) | 237
  Change at Month 30 | -1.378 (20.9437)
  Change at Month 54: number analyzed (Participants) | 42
  Change at Month 54 | -2.093 (19.5085)

13. Other Pre Specified Outcome: Change From Baseline in KCCQ Total Symptom Score at Months 12, 30 and 54: Cohort B
Description: KCCQ: 23-item, self-administered questionnaire that assesses health status and health-related quality of life in participants with heart failure. KCCQ quantifies 8 domains: physical limitations, symptom stability, symptom frequency, symptom burden, total symptom (mean of symptom frequency and symptom burden), self-efficacy, quality of life and social limitations). Scores were generated for each domain and scaled from 0 (worst) to 100 (best possible status). KCCQ Total Symptoms score was calculated as mean of the following domains- symptom frequency and symptom burden and transformed to a single score which ranged from 0 (worst) -100 (best possible status), higher scores = better health status. Data for change from baseline was reported as mean.
Time Frame: B3461045: Baseline (Day 1, pre-dose), Months 12, 30 and 54
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Cohort B: Tafamidis (Only in Extension Study)
Number analyzed (Participants) | 829
Units on a scale
  Change at Month 12 | 0.738 (19.1549)
  Change at Month 30: number analyzed (Participants) | 237
  Change at Month 30 | -1.112 (20.7952)
  Change at Month 54: number analyzed (Participants) | 42
  Change at Month 54 | -1.885 (19.4433)

14. Other Pre Specified Outcome: Number of Participants With Shift From Baseline in New York Heart Association (NYHA) Classification at Month 6, 12, 18, 24, 30, 36, 42, 48, 54 and 60
Description: NYHA classification: Class I: Participants with cardiovascular disease (CVD) but without resulting limitation of physical activity. Ordinary physical activity does not cause undue fatigue, palpitation, dyspnea, or anginal pain; Class II: Participants with CVD resulting in slight limitation of physical activity and were comfortable at rest. Ordinary physical activity results in fatigue, palpitation, dyspnea, or angina pain; Class III: participants with CVD resulting in marked limitation of physical activity and were comfortable at rest. Less than ordinary physical activity causes fatigue, palpitation, dyspnea, or anginal pain; Class IV: participants with CVD resulting in inability to carry on any physical activity without discomfort. Symptoms of cardiac insufficiency or of the anginal syndrome may be present even at rest. If any physical activity was undertaken, discomfort was increased.
Time Frame: B3461045: Baseline (Day 1, pre-dose), Months 6, 12, 18, 24, 30, 36, 42, 48, 54 and 60
Population: Safety analysis population included all participants (Cohorts A and B) who were enrolled in this study and taken at least 1 dose of study medication. All participants reported under "Number of Participants Analyzed" contributed data to the table; however, may not have evaluable data for every row. "Number Analyzed" signifies number of participants evaluable at specified time points. Therefore, this analysis (Cohort A) was based on the pooled dose groups, as per the SAP.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A: Tafamidis (Parent and Extension Study) | Cohort A: Placebo (Parent Study)/Tafamidis (Extension Study) | Cohort B: Tafamidis (Only in Extension Study)
Number analyzed (Participants) | 170 | 82 | 1476
Participants
  Month 6: number analyzed (Participants) | 155 | 66 | 1249
  Month 6: Class I (Baseline) to Class I | 13 | 4 | 132
  Month 6: Class I (Baseline) to Class II | 4 | 2 | 70
  Month 6: Class I (Baseline) to Class III | 0 | 0 | 8
  Month 6: Class I (Baseline) to Class IV | 0 | 0 | 0
  Month 6: Class II (Baseline) to Class I | 7 | 0 | 60
  Month 6: Class II (Baseline) to Class II | 65 | 20 | 542
  Month 6: Class II (Baseline) to Class III | 11 | 2 | 100
  Month 6: Class II (Baseline) to Class IV | 0 | 0 | 1
  Month 6: Class III (Baseline) to Class I | 1 | 0 | 4
  Month 6: Class III (Baseline) to Class II | 17 | 9 | 88
  Month 6: Class III (Baseline) to Class III | 34 | 24 | 226
  Month 6: Class III (Baseline) to Class IV | 0 | 0 | 2
  Month 6: Class IV (Baseline) to Class I | 0 | 0 | 1
  Month 6: Class IV (Baseline) to Class II | 1 | 1 | 2
  Month 6: Class IV (Baseline) to Class III | 1 | 3 | 10
  Month 6: Class IV (Baseline) to Class IV | 1 | 1 | 3
  Month 12: number analyzed (Participants) | 142 | 54 | 850
  Month 12: Class I (Baseline) to Class I | 10 | 4 | 94
  Month 12: Class I (Baseline) to Class II | 5 | 0 | 60
  Month 12: Class I (Baseline) to Class III | 1 | 0 | 3
  Month 12: Class I (Baseline) to Class IV | 0 | 0 | 0
  Month 12: Class II (Baseline) to Class I | 6 | 0 | 50
  Month 12: Class II (Baseline) to Class II | 63 | 16 | 371
  Month 12: Class II (Baseline) to Class III | 10 | 1 | 67
  Month 12: Class II (Baseline) to Class IV | 1 | 0 | 1
  Month 12: Class III (Baseline) to Class I | 3 | 0 | 1
  Month 12: Class III (Baseline) to Class II | 12 | 9 | 67
  Month 12: Class III (Baseline) to Class III | 31 | 23 | 127
  Month 12: Class III (Baseline) to Class IV | 0 | 0 | 0
  Month 12: Class IV (Baseline) to Class I | 0 | 0 | 0
  Month 12: Class IV (Baseline) to Class II | 0 | 0 | 1
  Month 12: Class IV (Baseline) to Class III | 0 | 1 | 7
  Month 12: Class IV (Baseline) to Class IV | 0 | 0 | 1
  Month 18: number analyzed (Participants) | 123 | 47 | 611
  Month 18: Class I (Baseline) to Class I | 5 | 4 | 64
  Month 18: Class I (Baseline) to Class II | 3 | 0 | 45
  Month 18: Class I (Baseline) to Class III | 0 | 0 | 3
  Month 18: Class I (Baseline) to Class IV | 0 | 0 | 0
  Month 18: Class II (Baseline) to Class I | 8 | 0 | 41
  Month 18: Class II (Baseline) to Class II | 49 | 15 | 259
  Month 18: Class II (Baseline) to Class III | 9 | 1 | 61
  Month 18: Class II (Baseline) to Class IV | 0 | 0 | 1
  Month 18: Class III (Baseline) to Class I | 2 | 0 | 5
  Month 18: Class III (Baseline) to Class II | 19 | 6 | 57
  Month 18: Class III (Baseline) to Class III | 24 | 19 | 70
  Month 18: Class III (Baseline) to Class IV | 0 | 0 | 0
  Month 18: Class IV (Baseline) to Class I | 2 | 0 | 0
  Month 18: Class IV (Baseline) to Class II | 0 | 0 | 2
  Month 18: Class IV (Baseline) to Class III | 2 | 2 | 3
  Month 18: Class IV (Baseline) to Class IV | 0 | 0 | 0
  Month 24: number analyzed (Participants) | 105 | 40 | 434
  Month 24: Class I (Baseline) to Class I | 4 | 4 | 42
  Month 24: Class I (Baseline) to Class II | 4 | 1 | 40
  Month 24: Class I (Baseline) to Class III | 2 | 1 | 0
  Month 24: Class I (Baseline) to Class IV | 0 | 0 | 0
  Month 24: Class II (Baseline) to Class I | 8 | 0 | 31
  Month 24: Class II (Baseline) to Class II | 49 | 12 | 191
  Month 24: Class II (Baseline) to Class III | 3 | 0 | 42
  Month 24: Class II (Baseline) to Class IV | 0 | 0 | 0
  Month 24: Class III (Baseline) to Class I | 4 | 0 | 3
  Month 24: Class III (Baseline) to Class II | 11 | 8 | 34
  Month 24: Class III (Baseline) to Class III | 17 | 14 | 46
  Month 24: Class III (Baseline) to Class IV | 0 | 0 | 0
  Month 24: Class IV (Baseline) to Class I | 0 | 0 | 0
  Month 24: Class IV (Baseline) to Class II | 1 | 0 | 1
  Month 24: Class IV (Baseline) to Class III | 2 | 0 | 4
  Month 24: Class IV (Baseline) to Class IV | 0 | 0 | 0
  Month 30: number analyzed (Participants) | 64 | 23 | 291
  Month 30: Class I (Baseline) to Class I | 1 | 1 | 27
  Month 30: Class I (Baseline) to Class II | 1 | 0 | 32
  Month 30: Class I (Baseline) to Class III | 0 | 0 | 1
  Month 30: Class I (Baseline) to Class IV | 0 | 0 | 0
  Month 30: Class II (Baseline) to Class I | 5 | 1 | 26
  Month 30: Class II (Baseline) to Class II | 27 | 7 | 129
  Month 30: Class II (Baseline) to Class III | 2 | 1 | 24
  Month 30: Class II (Baseline) to Class IV | 0 | 0 | 0
  Month 30: Class III (Baseline) to Class I | 4 | 0 | 2
  Month 30: Class III (Baseline) to Class II | 14 | 4 | 22
  Month 30: Class III (Baseline) to Class III | 10 | 9 | 24
  Month 30: Class III (Baseline) to Class IV | 0 | 0 | 0
  Month 30: Class IV (Baseline) to Class I | 0 | 0 | 0
  Month 30: Class IV (Baseline) to Class II | 0 | 0 | 2
  Month 30: Class IV (Baseline) to Class III | 0 | 0 | 2
  Month 30: Class IV (Baseline) to Class IV | 0 | 0 | 0
  Month 36: number analyzed (Participants) | 43 | 17 | 223
  Month 36: Class I (Baseline) to Class I | 1 | 2 | 21
  Month 36: Class I (Baseline) to Class II | 4 | 0 | 18
  Month 36: Class I (Baseline) to Class III | 0 | 0 | 0
  Month 36: Class I (Baseline) to Class IV | 0 | 0 | 0
  Month 36: Class II (Baseline) to Class I | 3 | 0 | 19
  Month 36: Class II (Baseline) to Class II | 19 | 7 | 101
  Month 36: Class II (Baseline) to Class III | 2 | 1 | 25
  Month 36: Class II (Baseline) to Class IV | 0 | 0 | 0
  Month 36: Class III (Baseline) to Class I | 1 | 0 | 3
  Month 36: Class III (Baseline) to Class II | 5 | 2 | 21
  Month 36: Class III (Baseline) to Class III | 7 | 4 | 14
  Month 36: Class III (Baseline) to Class IV | 0 | 0 | 0
  Month 36: Class IV (Baseline) to Class I | 0 | 0 | 0
  Month 36: Class IV (Baseline) to Class II | 1 | 0 | 1
  Month 36: Class IV (Baseline) to Class III | 0 | 1 | 0
  Month 36: Class IV (Baseline) to Class IV | 0 | 0 | 0
  Month 42: number analyzed (Participants) | 31 | 8 | 163
  Month 42: Class I (Baseline) to Class I | 0 | 0 | 16
  Month 42: Class I (Baseline) to Class II | 3 | 1 | 11
  Month 42: Class I (Baseline) to Class III | 0 | 0 | 1
  Month 42: Class I (Baseline) to Class IV | 0 | 0 | 0
  Month 42: Class II (Baseline) to Class I | 4 | 1 | 9
  Month 42: Class II (Baseline) to Class II | 14 | 4 | 77
  Month 42: Class II (Baseline) to Class III | 2 | 0 | 16
  Month 42: Class II (Baseline) to Class IV | 0 | 0 | 0
  Month 42: Class III (Baseline) to Class I | 1 | 0 | 1
  Month 42: Class III (Baseline) to Class II | 3 | 1 | 20
  Month 42: Class III (Baseline) to Class III | 4 | 1 | 12
  Month 42: Class III (Baseline) to Class IV | 0 | 0 | 0
  Month 42: Class IV (Baseline) to Class I | 0 | 0 | 0
  Month 42: Class IV (Baseline) to Class II | 0 | 0 | 0
  Month 42: Class IV (Baseline) to Class III | 0 | 0 | 0
  Month 42: Class IV (Baseline) to Class IV | 0 | 0 | 0
  Month 48: number analyzed (Participants) | 27 | 7 | 99
  Month 48: Class I (Baseline) to Class I | 0 | 0 | 6
  Month 48: Class I (Baseline) to Class II | 2 | 0 | 8
  Month 48: Class I (Baseline) to Class III | 0 | 0 | 0
  Month 48: Class I (Baseline) to Class IV | 0 | 0 | 0
  Month 48: Class II (Baseline) to Class I | 2 | 1 | 2
  Month 48: Class II (Baseline) to Class II | 12 | 4 | 54
  Month 48: Class II (Baseline) to Class III | 2 | 0 | 7
  Month 48: Class II (Baseline) to Class IV | 0 | 0 | 0
  Month 48: Class III (Baseline) to Class I | 2 | 0 | 0
  Month 48: Class III (Baseline) to Class II | 3 | 1 | 8
  Month 48: Class III (Baseline) to Class III | 4 | 1 | 13
  Month 48: Class III (Baseline) to Class IV | 0 | 0 | 0
  Month 48: Class IV (Baseline) to Class I | 0 | 0 | 0
  Month 48: Class IV (Baseline) to Class II | 0 | 0 | 0
  Month 48: Class IV (Baseline) to Class III | 0 | 0 | 1
  Month 48: Class IV (Baseline) to Class IV | 0 | 0 | 0
  Month 54: number analyzed (Participants) | 18 | 4 | 44
  Month 54: Class I (Baseline) to Class I | 0 | 0 | 1
  Month 54: Class I (Baseline) to Class II | 0 | 0 | 3
  Month 54: Class I (Baseline) to Class III | 0 | 0 | 0
  Month 54: Class I (Baseline) to Class IV | 0 | 0 | 0
  Month 54: Class II (Baseline) to Class I | 0 | 0 | 1
  Month 54: Class II (Baseline) to Class II | 7 | 3 | 22
  Month 54: Class II (Baseline) to Class III | 2 | 0 | 6
  Month 54: Class II (Baseline) to Class IV | 0 | 0 | 0
  Month 54: Class III (Baseline) to Class I | 3 | 0 | 0
  Month 54: Class III (Baseline) to Class II | 3 | 1 | 4
  Month 54: Class III (Baseline) to Class III | 3 | 0 | 7
  Month 54: Class III (Baseline) to Class IV | 0 | 0 | 0
  Month 54: Class IV (Baseline) to Class I | 0 | 0 | 0
  Month 54: Class IV (Baseline) to Class II | 0 | 0 | 0
  Month 54: Class IV (Baseline) to Class III | 0 | 0 | 0
  Month 54: Class IV (Baseline) to Class IV | 0 | 0 | 0
  Month 60: number analyzed (Participants) | 9 | 2 | 0
  Month 60: Class I (Baseline) to Class I | 0 | 0 |
  Month 60: Class I (Baseline) to Class II | 0 | 0 |
  Month 60: Class I (Baseline) to Class III | 0 | 0 |
  Month 60: Class I (Baseline) to Class IV | 0 | 0 |
  Month 60: Class II (Baseline) to Class I | 0 | 0 |
  Month 60: Class II (Baseline) to Class II | 4 | 0 |
  Month 60: Class II (Baseline) to Class III | 2 | 0 |
  Month 60: Class II (Baseline) to Class IV | 0 | 0 |
  Month 60: Class III (Baseline) to Class I | 1 | 0 |
  Month 60: Class III (Baseline) to Class II | 1 | 2 |
  Month 60: Class III (Baseline) to Class III | 1 | 0 |
  Month 60: Class III (Baseline) to Class IV | 0 | 0 |
  Month 60: Class IV (Baseline) to Class I | 0 | 0 |
  Month 60: Class IV (Baseline) to Class II | 0 | 0 |
  Month 60: Class IV (Baseline) to Class III | 0 | 0 |
  Month 60: Class IV (Baseline) to Class IV | 0 | 0 |

15. Other Pre Specified Outcome: Change From Baseline in Body Mass Index (BMI) at Months 6, 12, 18, 24, 30, 36, 42, 48, 54 and 60
Description: BMI was calculated as: body weight in kilogram (kg) divided by (/) square of body height measurement in meters square (m^2).
Time Frame: B3461045: Baseline (Day 1, pre-dose), Months 6, 12, 18, 24, 30, 36, 42, 48, 54 and 60
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: kg/m^2
Arm/Group | Cohort A: Tafamidis (Parent and Extension Study) | Cohort A: Placebo (Parent Study)/Tafamidis (Extension Study) | Cohort B: Tafamidis (Only in Extension Study)
Number analyzed (Participants) | 170 | 82 | 1476
kg/m^2
  Change at Month 6: number analyzed (Participants) | 155 | 67 | 1216
  Change at Month 6 | -0.07 (0.873) | -0.27 (0.900) | -0.24 (1.234)
  Change at Month 12: number analyzed (Participants) | 141 | 54 | 800
  Change at Month 12 | -0.21 (1.212) | -0.40 (1.440) | -0.20 (1.552)
  Change at Month 18: number analyzed (Participants) | 122 | 47 | 555
  Change at Month 18 | -0.38 (1.442) | -0.85 (1.502) | -0.30 (1.956)
  Change at Month 24: number analyzed (Participants) | 104 | 40 | 418
  Change at Month 24 | -0.36 (1.407) | -0.78 (1.668) | -0.43 (1.747)
  Change at Month 30: number analyzed (Participants) | 62 | 23 | 287
  Change at Month 30 | -0.71 (1.423) | -1.28 (1.814) | -0.41 (1.802)
  Change at Month 36: number analyzed (Participants) | 41 | 16 | 220
  Change at Month 36 | -1.18 (2.200) | -0.49 (1.852) | -0.69 (1.730)
  Change at Month 42: number analyzed (Participants) | 30 | 8 | 162
  Change at Month 42 | -0.91 (1.402) | -0.11 (1.523) | -0.74 (1.827)
  Change at Month 48: number analyzed (Participants) | 27 | 7 | 100
  Change at Month 48 | -1.14 (1.480) | -0.01 (1.927) | -0.83 (1.732)
  Change at Month 54: number analyzed (Participants) | 18 | 4 | 44
  Change at Month 54 | -1.03 (1.716) | -1.54 (0.528) | -1.24 (1.942)
  Change at Month 60: number analyzed (Participants) | 9 | 2 | 0
  Change at Month 60 | -0.93 (2.102) | -1.62 (0.834) |

16. Other Pre Specified Outcome: Change From Baseline in Modified Body Mass Index (mBMI) at Months 6, 12, 18, 24, 30, 36, 42, 48, 54 and 60
Description: Modified (m)BMI of participants was calculated to determine if there was any gastrointestinal involvement in participants. The mBMI was calculated by multiplying BMI by serum albumin concentration gram/liter (g/L).
Time Frame: B3461045: Baseline (Day 1, pre-dose), Months 6, 12, 18, 24, 30, 36, 42, 48, 54 and 60
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: (kg/m^2) *(g/L)
Arm/Group | Cohort A: Tafamidis (Parent and Extension Study) | Cohort A: Placebo (Parent Study)/Tafamidis (Extension Study) | Cohort B: Tafamidis (Only in Extension Study)
Number analyzed (Participants) | 170 | 82 | 1476
(kg/m^2) *(g/L)
  Change at Month 6: number analyzed (Participants) | 154 | 64 | 1037
  Change at Month 6 | -2.96 (36.046) | -10.91 (36.338) | -8.51 (51.329)
  Change at Month 12: number analyzed (Participants) | 140 | 51 | 674
  Change at Month 12 | -7.42 (49.840) | -16.09 (57.882) | -6.17 (66.094)
  Change at Month 18: number analyzed (Participants) | 121 | 44 | 455
  Change at Month 18 | -15.46 (60.361) | -35.46 (63.390) | -10.08 (85.605)
  Change at Month 24: number analyzed (Participants) | 104 | 38 | 345
  Change at Month 24 | -15.07 (58.706) | -32.33 (71.104) | -15.81 (74.009)
  Change at Month 30: number analyzed (Participants) | 62 | 22 | 234
  Change at Month 30 | -29.31 (61.003) | -52.81 (78.705) | -15.70 (79.724)
  Change at Month 36: number analyzed (Participants) | 41 | 15 | 172
  Change at Month 36 | -49.46 (98.257) | -17.81 (80.327) | -24.66 (74.366)
  Change at Month 42: number analyzed (Participants) | 30 | 7 | 135
  Change at Month 42 | -36.32 (58.130) | 1.59 (69.701) | -28.06 (78.987)
  Change at Month 48: number analyzed (Participants) | 27 | 6 | 87
  Change at Month 48 | -46.43 (62.394) | 14.05 (83.969) | -32.91 (71.745)
  Change at Month 54: number analyzed (Participants) | 18 | 3 | 36
  Change at Month 54 | -41.98 (74.883) | -52.80 (14.562) | -51.15 (79.618)
  Change at Month 60: number analyzed (Participants) | 9 | 1 | 0
  Change at Month 60 | -38.90 (92.253) | -41.20 (NA) — Standard deviation could not be calculated as only one participant was analyzed. |

17. Other Pre Specified Outcome: Change From Baseline in Troponin I Concentration at Months 6, 12, 18, 24, 30, 36, 42, 48, 54 and 60
Description: Troponin I is the cardiac markers. Higher level of the marker was indicative of heart damage. It was measure in nanogram per milliliter (ng/mL). Safety analysis population included all participants (Cohorts A and B) who were enrolled in this study and taken at least 1 dose of study medication.
Time Frame: B3461045: Baseline (Day 1, pre-dose), Months 6, 12, 18, 24, 30, 36, 42, 48, 54 and 60
Population: Analysis was performed using Safety analysis population."Number of Participants Analyzed"=number of participants evaluable.All participants reported under"Number of Participants Analyzed"contributed data to the table;however,may not have evaluable data for every row."Number Analyzed"=number of participants evaluable at specified time points.The measurement was not required for participants enrolled before Protocol Amendment4(PA-4).The analysis(Cohort A)was based on pooled dose groups,as per SAP.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Cohort A: Tafamidis (Parent and Extension Study) | Cohort A: Placebo (Parent Study)/Tafamidis (Extension Study) | Cohort B: Tafamidis (Only in Extension Study)
Number analyzed (Participants) | 170 | 82 | 495
ng/mL
  Change at Month 6: number analyzed (Participants) | 0 | 0 | 108
  Change at Month 6 |  |  | 0.012 (0.1706)
  Change at Month 12: number analyzed (Participants) | 165 | 81 | 99
  Change at Month 12 | 0.035 (0.3977) | 0.037 (0.0853) | 0.009 (0.0893)
  Change at Month 18: number analyzed (Participants) | 1 | 0 | 70
  Change at Month 18 | 0.040 (NA) — Standard deviation could not be calculated as only one participant was analyzed. |  | -0.007 (0.0786)
  Change at Month 24: number analyzed (Participants) | 2 | 3 | 64
  Change at Month 24 | 0.000 (0.0566) | 0.033 (0.0306) | -0.031 (0.2031)
  Change at Month 30: number analyzed (Participants) | 168 | 80 | 64
  Change at Month 30 | 0.022 (0.1599) | 0.100 (0.1728) | -0.033 (0.2055)
  Change at Month 36: number analyzed (Participants) | 27 | 11 | 64
  Change at Month 36 | 0.009 (0.0579) | 0.018 (0.1057) | -0.034 (0.1913)
  Change at Month 42: number analyzed (Participants) | 26 | 6 | 24
  Change at Month 42 | -0.002 (0.0795) | -0.047 (0.0755) | -0.021 (0.2484)
  Change at Month 48: number analyzed (Participants) | 26 | 6 | 2
  Change at Month 48 | 0.016 (0.0795) | -0.067 (0.2040) | -0.100 (0.0000)
  Change at Month 54: number analyzed (Participants) | 14 | 3 | 0
  Change at Month 54 | -0.033 (0.0792) | -0.363 (0.6080) |
  Change at Month 60: number analyzed (Participants) | 8 | 2 | 0
  Change at Month 60 | -0.040 (0.0414) | 0.035 (0.0354) |

18. Other Pre Specified Outcome: Change From Baseline in N-Terminal Prohormone Brain Natriuretic Peptide (NT-proBNP) Concentration at Months 6, 12, 18, 24, 30, 36, 42, 48, 54 and 60
Description: NT-proBNP was a cardiac marker which had the prognostic value for participants with heart failure or left ventricular dysfunction. It was measure in picomole per liter (pmole/L). Higher level of the marker was indicative of heart damage. Safety analysis population included all participants (Cohorts A and B) who were enrolled in this study and taken at least 1 dose of study medication.
Time Frame: B3461045: Baseline (Day 1, pre-dose), Months 6, 12, 18, 24, 30, 36, 42, 48, 54 and 60
Population: Analysis was performed using Safety analysis population. "Number of Participants Analyzed"= number of participants evaluable. All participants reported under "Number of Participants Analyzed" contributed data to the table; however, may not have evaluable data for every row. "Number Analyzed"= number of participants evaluable at specified time points. This measurement was not required for participants enrolled before PA-4. This analysis (Cohort A) was based on pooled dose groups, as per SAP.
Measure: Mean (Standard Deviation); unit: pmole/L
Arm/Group | Cohort A: Tafamidis (Parent and Extension Study) | Cohort A: Placebo (Parent Study)/Tafamidis (Extension Study) | Cohort B: Tafamidis (Only in Extension Study)
Number analyzed (Participants) | 170 | 82 | 516
pmole/L
  Change at Month 6: number analyzed (Participants) | 0 | 0 | 108
  Change at Month 6 |  |  | 24.820 (171.2075)
  Change at Month 12: number analyzed (Participants) | 167 | 80 | 101
  Change at Month 12 | 31.117 (220.9279) | 127.973 (226.7727) | 32.686 (180.4921)
  Change at Month 18: number analyzed (Participants) | 1 | 0 | 79
  Change at Month 18 | 226.442 (NA) — Standard deviation could not be calculated as only one participant was analyzed. |  | 71.582 (329.5411)
  Change at Month 24: number analyzed (Participants) | 2 | 3 | 69
  Change at Month 24 | 131.334 (119.5258) | 256.442 (101.8073) | 92.899 (320.6054)
  Change at Month 30: number analyzed (Participants) | 170 | 81 | 70
  Change at Month 30 | 159.596 (404.8483) | 417.682 (597.9224) | 149.049 (320.8814)
  Change at Month 36: number analyzed (Participants) | 29 | 11 | 63
  Change at Month 36 | 322.963 (215.1605) | 420.196 (251.8446) | 88.895 (227.7375)
  Change at Month 42: number analyzed (Participants) | 26 | 6 | 24
  Change at Month 42 | 419.034 (315.6436) | 324.211 (173.6652) | 191.318 (482.3582)
  Change at Month 48: number analyzed (Participants) | 26 | 6 | 2
  Change at Month 48 | 492.154 (387.4700) | 400.571 (228.4343) | 264.566 (78.7059)
  Change at Month 54: number analyzed (Participants) | 17 | 3 | 0
  Change at Month 54 | 405.887 (457.6349) | 340.082 (190.6412) |
  Change at Month 60: number analyzed (Participants) | 9 | 2 | 0
  Change at Month 60 | 392.363 (271.2883) | 314.184 (274.6756) |

ADVERSE EVENTS:
Time Frame: B3461045: From first dose of treatment up to 28 days post last dose of study treatment (approximately up to 61 months)
Description: Same event may appear as non-SAE and SAE, what is presented are distinct events. Event may be categorized as serious in 1 participant and as non-serious in another participant or 1 participant may have experienced both serious and non-serious event during study. Safety analysis population consisted of all participants (Cohorts A and B) who were enrolled in this study and taken at least 1 dose of study medication.
Arm/Group | Cohort A: Tafamidis (Parent and Extension Study) | Cohort A: Placebo (Parent Study)/Tafamidis (Extension Study) | Cohort B: Tafamidis (Only in Extension Study)
All-Cause Mortality (participants affected / at risk) | 45/170 | 33/82 | 203/1476
Serious Adverse Events (participants affected / at risk) | 132/170 | 64/82 | 736/1476
Other Adverse Events (participants affected / at risk) | 152/170 | 76/82 | 1023/1476
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort A: Tafamidis (Parent and Extension Study) (N=170) | Cohort A: Placebo (Parent Study)/Tafamidis (Extension Study) (N=82) | Cohort B: Tafamidis (Only in Extension Study) (N=1476)
Anaemia (Blood and lymphatic system disorders) | 2 | 0 | 17
Aplastic anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1
Blood loss anaemia (Blood and lymphatic system disorders) | 1 | 0 | 2
Coagulopathy (Blood and lymphatic system disorders) | 0 | 0 | 1
Deficiency anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1
Immune thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 2
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 | 0 | 2
Leukocytosis (Blood and lymphatic system disorders) | 0 | 0 | 1
Normochromic normocytic anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1
Spontaneous haematoma (Blood and lymphatic system disorders) | 1 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0 | 0
Acute coronary syndrome (Cardiac disorders) | 0 | 0 | 2
Acute left ventricular failure (Cardiac disorders) | 2 | 3 | 7
Acute myocardial infarction (Cardiac disorders) | 2 | 2 | 7
Angina pectoris (Cardiac disorders) | 2 | 0 | 11
Angina unstable (Cardiac disorders) | 1 | 0 | 0
Aortic valve stenosis (Cardiac disorders) | 0 | 1 | 2
Arrhythmia (Cardiac disorders) | 3 | 0 | 2
Arrhythmia supraventricular (Cardiac disorders) | 0 | 0 | 2
Atrial fibrillation (Cardiac disorders) | 11 | 8 | 62
Atrial flutter (Cardiac disorders) | 4 | 1 | 18
Atrial tachycardia (Cardiac disorders) | 0 | 1 | 4
Atrioventricular block (Cardiac disorders) | 4 | 1 | 8
Atrioventricular block complete (Cardiac disorders) | 1 | 0 | 16
Bifascicular block (Cardiac disorders) | 0 | 0 | 1
Bradyarrhythmia (Cardiac disorders) | 1 | 0 | 1
Bradycardia (Cardiac disorders) | 2 | 2 | 11
Bundle branch block bilateral (Cardiac disorders) | 0 | 0 | 1
Bundle branch block left (Cardiac disorders) | 0 | 0 | 4
Bundle branch block right (Cardiac disorders) | 0 | 0 | 2
Cardiac amyloidosis (Cardiac disorders) | 2 | 2 | 16
Cardiac arrest (Cardiac disorders) | 6 | 3 | 14
Cardiac failure (Cardiac disorders) | 30 | 17 | 169
Cardiac failure acute (Cardiac disorders) | 13 | 10 | 48
Cardiac failure chronic (Cardiac disorders) | 1 | 4 | 10
Cardiac failure congestive (Cardiac disorders) | 17 | 14 | 52
Cardiac flutter (Cardiac disorders) | 1 | 0 | 0
Cardio-respiratory arrest (Cardiac disorders) | 0 | 1 | 0
Cardio-respiratory distress (Cardiac disorders) | 0 | 0 | 1
Cardiogenic shock (Cardiac disorders) | 3 | 2 | 20
Cardiomyopathy (Cardiac disorders) | 1 | 0 | 0
Cardiopulmonary failure (Cardiac disorders) | 0 | 2 | 0
Cardiorenal syndrome (Cardiac disorders) | 0 | 0 | 3
Cardiovascular insufficiency (Cardiac disorders) | 0 | 0 | 1
Chronic left ventricular failure (Cardiac disorders) | 1 | 3 | 3
Conduction disorder (Cardiac disorders) | 0 | 0 | 5
Coronary artery disease (Cardiac disorders) | 1 | 0 | 1
Coronary artery embolism (Cardiac disorders) | 1 | 0 | 0
Coronary artery stenosis (Cardiac disorders) | 0 | 0 | 1
Left ventricular dysfunction (Cardiac disorders) | 0 | 0 | 1
Left ventricular failure (Cardiac disorders) | 1 | 1 | 6
Low cardiac output syndrome (Cardiac disorders) | 0 | 1 | 1
Mitral valve incompetence (Cardiac disorders) | 1 | 0 | 0
Myocardial infarction (Cardiac disorders) | 1 | 0 | 3
Myocardial ischaemia (Cardiac disorders) | 0 | 0 | 1
Nodal arrhythmia (Cardiac disorders) | 0 | 0 | 1
Nodal rhythm (Cardiac disorders) | 0 | 0 | 1
Palpitations (Cardiac disorders) | 0 | 0 | 1
Paroxysmal atrioventricular block (Cardiac disorders) | 0 | 0 | 1
Pericardial effusion (Cardiac disorders) | 3 | 1 | 2
Pericarditis (Cardiac disorders) | 0 | 0 | 1
Restrictive cardiomyopathy (Cardiac disorders) | 0 | 0 | 1
Right ventricular dysfunction (Cardiac disorders) | 0 | 0 | 1
Right ventricular failure (Cardiac disorders) | 0 | 1 | 0
Sinoatrial block (Cardiac disorders) | 0 | 0 | 1
Sinus arrest (Cardiac disorders) | 1 | 0 | 0
Sinus node dysfunction (Cardiac disorders) | 1 | 1 | 10
Supraventricular tachycardia (Cardiac disorders) | 0 | 0 | 7
Tachyarrhythmia (Cardiac disorders) | 0 | 1 | 0
Tachycardia (Cardiac disorders) | 1 | 0 | 0
Torsade de pointes (Cardiac disorders) | 0 | 1 | 0
Tricuspid valve incompetence (Cardiac disorders) | 0 | 0 | 2
Ventricular arrhythmia (Cardiac disorders) | 1 | 0 | 0
Ventricular dysfunction (Cardiac disorders) | 0 | 0 | 4
Ventricular fibrillation (Cardiac disorders) | 1 | 0 | 1
Ventricular tachycardia (Cardiac disorders) | 3 | 6 | 17
Familial amyloidosis (Congenital, familial and genetic disorders) | 4 | 1 | 10
Hereditary neuropathic amyloidosis (Congenital, familial and genetic disorders) | 0 | 0 | 2
Meniere's disease (Ear and labyrinth disorders) | 0 | 0 | 1
Vertigo (Ear and labyrinth disorders) | 1 | 0 | 1
Hyperthyroidism (Endocrine disorders) | 0 | 0 | 2
Amaurosis fugax (Eye disorders) | 0 | 0 | 1
Blindness unilateral (Eye disorders) | 0 | 0 | 1
Cataract (Eye disorders) | 1 | 0 | 0
Charles Bonnet syndrome (Eye disorders) | 1 | 0 | 0
Optic ischaemic neuropathy (Eye disorders) | 0 | 0 | 1
Orbital haematoma (Eye disorders) | 0 | 0 | 1
Retinal detachment (Eye disorders) | 0 | 0 | 1
Vision blurred (Eye disorders) | 1 | 0 | 0
Vitreous haemorrhage (Eye disorders) | 1 | 0 | 0
Abdominal adhesions (Gastrointestinal disorders) | 1 | 0 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 1
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 6
Abdominal pain lower (Gastrointestinal disorders) | 0 | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 2 | 0 | 0
Acute abdomen (Gastrointestinal disorders) | 0 | 0 | 1
Appendiceal mucocoele (Gastrointestinal disorders) | 0 | 0 | 1
Ascites (Gastrointestinal disorders) | 2 | 1 | 8
Chronic gastritis (Gastrointestinal disorders) | 1 | 0 | 0
Colitis (Gastrointestinal disorders) | 0 | 0 | 1
Colitis microscopic (Gastrointestinal disorders) | 0 | 0 | 1
Constipation (Gastrointestinal disorders) | 2 | 2 | 2
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 2
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 2
Faecaloma (Gastrointestinal disorders) | 2 | 1 | 0
Gastric ulcer (Gastrointestinal disorders) | 1 | 0 | 1
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1
Gastritis (Gastrointestinal disorders) | 0 | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 4 | 1 | 13
Gastrointestinal ulcer haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1
Gastrointestinal vascular malformation haemorrhagic (Gastrointestinal disorders) | 0 | 0 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 1
Haemorrhoids (Gastrointestinal disorders) | 0 | 0 | 1
Ileus (Gastrointestinal disorders) | 0 | 0 | 1
Impaired gastric emptying (Gastrointestinal disorders) | 0 | 1 | 1
Incarcerated inguinal hernia (Gastrointestinal disorders) | 1 | 0 | 0
Incarcerated umbilical hernia (Gastrointestinal disorders) | 0 | 1 | 0
Inguinal hernia (Gastrointestinal disorders) | 0 | 2 | 4
Inguinal hernia strangulated (Gastrointestinal disorders) | 0 | 0 | 1
Intestinal ischaemia (Gastrointestinal disorders) | 0 | 0 | 1
Intestinal obstruction (Gastrointestinal disorders) | 1 | 1 | 3
Intra-abdominal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1
Large intestine perforation (Gastrointestinal disorders) | 0 | 0 | 1
Large intestine polyp (Gastrointestinal disorders) | 0 | 0 | 1
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1
Melaena (Gastrointestinal disorders) | 1 | 0 | 4
Mesenteric vascular insufficiency (Gastrointestinal disorders) | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 1 | 3
Oesophageal motility disorder (Gastrointestinal disorders) | 0 | 0 | 1
Oesophageal ulcer (Gastrointestinal disorders) | 1 | 0 | 1
Pancreatitis (Gastrointestinal disorders) | 0 | 0 | 2
Pancreatitis acute (Gastrointestinal disorders) | 0 | 0 | 2
Pneumoperitoneum (Gastrointestinal disorders) | 1 | 0 | 0
Portal hypertensive gastropathy (Gastrointestinal disorders) | 0 | 0 | 1
Rectal haemorrhage (Gastrointestinal disorders) | 3 | 0 | 7
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 1 | 4
Umbilical hernia (Gastrointestinal disorders) | 1 | 1 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 6
Vomiting (Gastrointestinal disorders) | 1 | 1 | 4
Asthenia (General disorders) | 2 | 2 | 5
Chest pain (General disorders) | 4 | 0 | 5
Death (General disorders) | 0 | 1 | 7
Discomfort (General disorders) | 1 | 0 | 0
Disease progression (General disorders) | 4 | 3 | 22
Fatigue (General disorders) | 1 | 0 | 3
General physical health deterioration (General disorders) | 1 | 1 | 11
Generalised oedema (General disorders) | 1 | 0 | 3
Hernia (General disorders) | 0 | 0 | 1
Hypothermia (General disorders) | 1 | 0 | 0
Implant site haematoma (General disorders) | 0 | 0 | 1
Inflammation (General disorders) | 0 | 0 | 1
Multi-organ disorder (General disorders) | 0 | 0 | 1
Multiple organ dysfunction syndrome (General disorders) | 1 | 0 | 1
Non-cardiac chest pain (General disorders) | 1 | 0 | 0
Oedema peripheral (General disorders) | 0 | 0 | 6
Pain (General disorders) | 0 | 1 | 2
Peripheral swelling (General disorders) | 0 | 0 | 1
Pyrexia (General disorders) | 0 | 0 | 3
Sudden death (General disorders) | 0 | 0 | 6
Systemic inflammatory response syndrome (General disorders) | 2 | 0 | 0
Biliary colic (Hepatobiliary disorders) | 0 | 0 | 1
Cardiac cirrhosis (Hepatobiliary disorders) | 0 | 0 | 1
Cholangitis (Hepatobiliary disorders) | 0 | 0 | 2
Cholecystitis acute (Hepatobiliary disorders) | 0 | 0 | 5
Congestive hepatopathy (Hepatobiliary disorders) | 1 | 1 | 1
Hepatic cirrhosis (Hepatobiliary disorders) | 2 | 0 | 1
Hepatic failure (Hepatobiliary disorders) | 0 | 0 | 3
Hepatic function abnormal (Hepatobiliary disorders) | 0 | 0 | 1
Hepatitis acute (Hepatobiliary disorders) | 0 | 0 | 1
Hepatomegaly (Hepatobiliary disorders) | 0 | 0 | 1
Ischaemic hepatitis (Hepatobiliary disorders) | 0 | 0 | 1
Jaundice (Hepatobiliary disorders) | 0 | 0 | 1
Acquired ATTR amyloidosis (Immune system disorders) | 0 | 0 | 1
Amyloidosis (Immune system disorders) | 0 | 0 | 2
Anaphylactic reaction (Immune system disorders) | 0 | 0 | 1
Graft versus host disease (Immune system disorders) | 0 | 0 | 1
Primary amyloidosis (Immune system disorders) | 0 | 0 | 1
Abscess limb (Infections and infestations) | 0 | 1 | 1
Appendicitis (Infections and infestations) | 0 | 0 | 2
Arthritis bacterial (Infections and infestations) | 1 | 0 | 3
Arthritis infective (Infections and infestations) | 0 | 0 | 2
Bacteraemia (Infections and infestations) | 0 | 1 | 4
Bacterial pyelonephritis (Infections and infestations) | 0 | 0 | 1
Beta haemolytic streptococcal infection (Infections and infestations) | 0 | 0 | 1
Bronchitis (Infections and infestations) | 0 | 1 | 2
Bronchitis viral (Infections and infestations) | 1 | 0 | 0
Bursitis infective (Infections and infestations) | 0 | 0 | 2
COVID-19 (Infections and infestations) | 2 | 1 | 16
COVID-19 pneumonia (Infections and infestations) | 1 | 1 | 9
Cardiac infection (Infections and infestations) | 0 | 0 | 1
Cellulitis (Infections and infestations) | 8 | 5 | 18
Cellulitis staphylococcal (Infections and infestations) | 1 | 0 | 0
Device related infection (Infections and infestations) | 1 | 1 | 0
Diabetic foot infection (Infections and infestations) | 0 | 0 | 1
Diverticulitis (Infections and infestations) | 0 | 0 | 5
Diverticulitis intestinal perforated (Infections and infestations) | 0 | 0 | 1
Endocarditis (Infections and infestations) | 0 | 0 | 1
Endophthalmitis (Infections and infestations) | 0 | 0 | 1
Erysipelas (Infections and infestations) | 1 | 1 | 4
Escherichia sepsis (Infections and infestations) | 2 | 0 | 0
Extradural abscess (Infections and infestations) | 0 | 1 | 0
Gastroenteritis (Infections and infestations) | 0 | 1 | 1
Gastrointestinal viral infection (Infections and infestations) | 0 | 0 | 1
Haematoma infection (Infections and infestations) | 0 | 0 | 1
Hepatitis A (Infections and infestations) | 0 | 0 | 1
Herpes zoster (Infections and infestations) | 1 | 0 | 0
Herpes zoster meningoencephalitis (Infections and infestations) | 0 | 0 | 1
Herpes zoster meningomyelitis (Infections and infestations) | 0 | 0 | 1
Implant site infection (Infections and infestations) | 1 | 1 | 0
Infection (Infections and infestations) | 0 | 0 | 2
Infectious pleural effusion (Infections and infestations) | 0 | 0 | 1
Infective exacerbation of chronic obstructive airways disease (Infections and infestations) | 0 | 0 | 1
Influenza (Infections and infestations) | 1 | 1 | 2
Legionella infection (Infections and infestations) | 0 | 0 | 1
Localised infection (Infections and infestations) | 0 | 1 | 0
Lower respiratory tract infection (Infections and infestations) | 0 | 0 | 2
Meningitis (Infections and infestations) | 0 | 0 | 1
Meningitis bacterial (Infections and infestations) | 0 | 0 | 1
Necrotising fasciitis (Infections and infestations) | 0 | 0 | 1
Oesophageal candidiasis (Infections and infestations) | 0 | 1 | 0
Osteomyelitis (Infections and infestations) | 1 | 0 | 0
Pericarditis infective (Infections and infestations) | 0 | 0 | 1
Peritonitis (Infections and infestations) | 0 | 0 | 2
Peritonsillar abscess (Infections and infestations) | 1 | 0 | 0
Pneumonia (Infections and infestations) | 12 | 9 | 39
Pneumonia aspiration (Infections and infestations) | 1 | 1 | 5
Pneumonia bacterial (Infections and infestations) | 1 | 0 | 3
Pneumonia klebsiella (Infections and infestations) | 0 | 0 | 1
Pneumonia pneumococcal (Infections and infestations) | 2 | 0 | 0
Pneumonia staphylococcal (Infections and infestations) | 1 | 0 | 0
Pneumonia streptococcal (Infections and infestations) | 1 | 0 | 0
Pneumonia viral (Infections and infestations) | 0 | 0 | 1
Post procedural sepsis (Infections and infestations) | 0 | 0 | 2
Pseudomonal sepsis (Infections and infestations) | 0 | 0 | 1
Pulmonary sepsis (Infections and infestations) | 0 | 0 | 1
Pyelonephritis (Infections and infestations) | 1 | 0 | 0
Respiratory moniliasis (Infections and infestations) | 0 | 0 | 1
Respiratory tract infection (Infections and infestations) | 0 | 0 | 7
Respiratory tract infection bacterial (Infections and infestations) | 0 | 0 | 1
Scrotal cellulitis (Infections and infestations) | 0 | 0 | 1
Sepsis (Infections and infestations) | 8 | 4 | 17
Septic shock (Infections and infestations) | 1 | 1 | 10
Sialoadenitis (Infections and infestations) | 0 | 0 | 1
Spontaneous bacterial peritonitis (Infections and infestations) | 0 | 0 | 3
Staphylococcal bacteraemia (Infections and infestations) | 0 | 0 | 3
Staphylococcal infection (Infections and infestations) | 1 | 0 | 0
Staphylococcal sepsis (Infections and infestations) | 0 | 0 | 1
Streptococcal bacteraemia (Infections and infestations) | 0 | 0 | 1
Streptococcal sepsis (Infections and infestations) | 0 | 0 | 1
Superinfection fungal (Infections and infestations) | 0 | 0 | 1
Tracheobronchitis (Infections and infestations) | 0 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 1
Urinary tract infection (Infections and infestations) | 2 | 0 | 17
Urosepsis (Infections and infestations) | 1 | 1 | 5
Vascular device infection (Infections and infestations) | 0 | 0 | 1
Viral infection (Infections and infestations) | 1 | 0 | 0
Acetabulum fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Cardiac procedure complication (Injury, poisoning and procedural complications) | 1 | 0 | 0
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 0 | 0 | 2
Chest injury (Injury, poisoning and procedural complications) | 0 | 1 | 1
Clavicle fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Complications of transplanted kidney (Injury, poisoning and procedural complications) | 1 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 1
Craniocerebral injury (Injury, poisoning and procedural complications) | 1 | 0 | 1
Craniofacial fracture (Injury, poisoning and procedural complications) | 1 | 0 | 1
Fall (Injury, poisoning and procedural complications) | 10 | 5 | 25
Fat embolism (Injury, poisoning and procedural complications) | 0 | 0 | 1
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 | 1 | 2
Femur fracture (Injury, poisoning and procedural complications) | 2 | 1 | 4
Foot fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Head injury (Injury, poisoning and procedural complications) | 1 | 1 | 3
Hip fracture (Injury, poisoning and procedural complications) | 0 | 0 | 9
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 0 | 3
Ilium fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Injury (Injury, poisoning and procedural complications) | 0 | 0 | 1
Joint dislocation (Injury, poisoning and procedural complications) | 1 | 0 | 0
Limb injury (Injury, poisoning and procedural complications) | 1 | 0 | 3
Meniscus injury (Injury, poisoning and procedural complications) | 1 | 0 | 0
Muscle strain (Injury, poisoning and procedural complications) | 1 | 0 | 0
Nasal injury (Injury, poisoning and procedural complications) | 0 | 0 | 1
Overdose (Injury, poisoning and procedural complications) | 0 | 0 | 1
Pelvic fracture (Injury, poisoning and procedural complications) | 0 | 1 | 4
Periprosthetic fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Periprosthetic osteolysis (Injury, poisoning and procedural complications) | 0 | 0 | 1
Post procedural constipation (Injury, poisoning and procedural complications) | 0 | 0 | 1
Post procedural haematoma (Injury, poisoning and procedural complications) | 0 | 0 | 1
Post procedural haematuria (Injury, poisoning and procedural complications) | 0 | 0 | 1
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 | 0 | 3
Procedural complication (Injury, poisoning and procedural complications) | 1 | 0 | 0
Procedural pneumothorax (Injury, poisoning and procedural complications) | 1 | 0 | 0
Pulmonary contusion (Injury, poisoning and procedural complications) | 0 | 0 | 1
Radius fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Rib fracture (Injury, poisoning and procedural complications) | 1 | 0 | 4
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 0 | 3
Seroma (Injury, poisoning and procedural complications) | 0 | 0 | 1
Skin abrasion (Injury, poisoning and procedural complications) | 0 | 1 | 1
Skin laceration (Injury, poisoning and procedural complications) | 0 | 0 | 2
Spinal compression fracture (Injury, poisoning and procedural complications) | 3 | 1 | 1
Spinal fracture (Injury, poisoning and procedural complications) | 0 | 0 | 2
Splenic injury (Injury, poisoning and procedural complications) | 0 | 0 | 1
Splenic rupture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Sternal fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Subdural haematoma (Injury, poisoning and procedural complications) | 1 | 0 | 10
Tendon rupture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Toxicity to various agents (Injury, poisoning and procedural complications) | 1 | 0 | 0
Traumatic intracranial haemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 1
Urinary tract stoma complication (Injury, poisoning and procedural complications) | 0 | 0 | 1
Vasoplegia syndrome (Injury, poisoning and procedural complications) | 0 | 0 | 1
Wound haemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 1
Wound secretion (Injury, poisoning and procedural complications) | 0 | 0 | 1
Wrist fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Activated partial thromboplastin time prolonged (Investigations) | 0 | 0 | 1
Anticoagulation drug level above therapeutic (Investigations) | 1 | 1 | 0
Apnoea test (Investigations) | 0 | 0 | 1
Blood bilirubin increased (Investigations) | 0 | 0 | 1
Blood potassium abnormal (Investigations) | 0 | 1 | 0
Blood urea increased (Investigations) | 0 | 1 | 0
Bronchial aspiration procedure (Investigations) | 0 | 0 | 1
Ejection fraction (Investigations) | 0 | 0 | 1
Ejection fraction decreased (Investigations) | 0 | 0 | 1
Haemoglobin decreased (Investigations) | 0 | 1 | 0
Heart rate irregular (Investigations) | 0 | 0 | 1
International normalised ratio increased (Investigations) | 0 | 0 | 1
Peritoneal fluid analysis (Investigations) | 0 | 1 | 0
SARS-CoV-2 test positive (Investigations) | 0 | 0 | 4
Troponin increased (Investigations) | 0 | 0 | 3
Cachexia (Metabolism and nutrition disorders) | 0 | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0 | 2
Dehydration (Metabolism and nutrition disorders) | 0 | 5 | 7
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 0 | 1
Diabetic metabolic decompensation (Metabolism and nutrition disorders) | 0 | 0 | 1
Electrolyte imbalance (Metabolism and nutrition disorders) | 0 | 1 | 0
Failure to thrive (Metabolism and nutrition disorders) | 0 | 0 | 4
Fluid retention (Metabolism and nutrition disorders) | 0 | 0 | 2
Gout (Metabolism and nutrition disorders) | 1 | 0 | 9
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Hyperglycaemic hyperosmolar nonketotic syndrome (Metabolism and nutrition disorders) | 0 | 0 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 2 | 1 | 8
Hypernatraemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Hypervolaemia (Metabolism and nutrition disorders) | 0 | 2 | 8
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 2
Hypokalaemia (Metabolism and nutrition disorders) | 2 | 2 | 9
Hyponatraemia (Metabolism and nutrition disorders) | 3 | 1 | 4
Hypovolaemia (Metabolism and nutrition disorders) | 0 | 1 | 2
Malnutrition (Metabolism and nutrition disorders) | 0 | 0 | 1
Metabolic alkalosis (Metabolism and nutrition disorders) | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 9
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 0 | 4
Chondrocalcinosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Dupuytren's contracture (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Gouty arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2
Greater trochanteric pain syndrome (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Haemarthrosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 3
Haematoma muscle (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Immunoglobulin G4 related disease (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 4
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 2 | 0 | 9
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2
Pathological fracture (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 4
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Tenosynovitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 4
Adrenal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Anal squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 2 | 9
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 1
Bladder transitional cell carcinoma recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Bowen's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Central nervous system melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Chronic myelomonocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Colon neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Diffuse large B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Hormone-dependent prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Metastases to lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Myelodysplastic syndrome with excess blasts (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Neuroendocrine carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Neuroendocrine tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Non-Hodgkin's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Non-small cell lung cancer stage IIIB (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Oesophageal squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Oncocytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Primary pulmonary melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 0 | 5
Prostate cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 1
Renal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 2
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 6
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 4
Ataxia (Nervous system disorders) | 0 | 0 | 1
Brain compression (Nervous system disorders) | 1 | 0 | 0
Brain injury (Nervous system disorders) | 2 | 0 | 0
Carpal tunnel syndrome (Nervous system disorders) | 0 | 0 | 1
Cerebral artery embolism (Nervous system disorders) | 0 | 0 | 1
Cerebral haemorrhage (Nervous system disorders) | 0 | 0 | 1
Cerebral infarction (Nervous system disorders) | 1 | 0 | 0
Cerebral ischaemia (Nervous system disorders) | 2 | 0 | 0
Cerebrospinal fluid leakage (Nervous system disorders) | 0 | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 2 | 3 | 17
Cervical radiculopathy (Nervous system disorders) | 0 | 0 | 1
Cognitive disorder (Nervous system disorders) | 0 | 0 | 6
Coma (Nervous system disorders) | 1 | 0 | 0
Dementia (Nervous system disorders) | 3 | 1 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 5
Dysarthria (Nervous system disorders) | 0 | 1 | 1
Embolic stroke (Nervous system disorders) | 1 | 0 | 0
Encephalopathy (Nervous system disorders) | 3 | 0 | 3
Epilepsy (Nervous system disorders) | 0 | 0 | 1
Haemorrhage intracranial (Nervous system disorders) | 0 | 0 | 1
Haemorrhagic transformation stroke (Nervous system disorders) | 0 | 0 | 1
Headache (Nervous system disorders) | 1 | 0 | 0
Hemianopia (Nervous system disorders) | 1 | 0 | 0
Hemianopia homonymous (Nervous system disorders) | 0 | 0 | 1
Hepatic encephalopathy (Nervous system disorders) | 2 | 0 | 1
Ischaemic cerebral infarction (Nervous system disorders) | 0 | 0 | 1
Ischaemic stroke (Nervous system disorders) | 1 | 3 | 11
Lethargy (Nervous system disorders) | 0 | 0 | 1
Loss of consciousness (Nervous system disorders) | 2 | 0 | 1
Metabolic encephalopathy (Nervous system disorders) | 1 | 0 | 1
Neuralgia (Nervous system disorders) | 0 | 0 | 1
Neuropathy peripheral (Nervous system disorders) | 0 | 0 | 1
Peripheral sensorimotor neuropathy (Nervous system disorders) | 0 | 0 | 1
Polyneuropathy (Nervous system disorders) | 1 | 0 | 1
Presyncope (Nervous system disorders) | 0 | 0 | 4
Radiculopathy (Nervous system disorders) | 0 | 0 | 1
Seizure (Nervous system disorders) | 0 | 0 | 1
Somnolence (Nervous system disorders) | 1 | 0 | 1
Subarachnoid haemorrhage (Nervous system disorders) | 0 | 1 | 0
Syncope (Nervous system disorders) | 6 | 2 | 42
Transient global amnesia (Nervous system disorders) | 0 | 0 | 1
Transient ischaemic attack (Nervous system disorders) | 0 | 0 | 9
Uraemic encephalopathy (Nervous system disorders) | 0 | 0 | 1
Vascular dementia (Nervous system disorders) | 0 | 0 | 1
Vascular encephalopathy (Nervous system disorders) | 0 | 1 | 0
Device capturing issue (Product Issues) | 1 | 0 | 0
Device dislocation (Product Issues) | 0 | 0 | 1
Device failure (Product Issues) | 0 | 0 | 1
Device inappropriate shock delivery (Product Issues) | 1 | 0 | 0
Device loosening (Product Issues) | 0 | 0 | 1
Device malfunction (Product Issues) | 2 | 0 | 1
Device occlusion (Product Issues) | 0 | 0 | 1
Agitation (Psychiatric disorders) | 0 | 0 | 1
Anxiety (Psychiatric disorders) | 0 | 0 | 1
Completed suicide (Psychiatric disorders) | 1 | 0 | 0
Confusional state (Psychiatric disorders) | 0 | 0 | 6
Delirium (Psychiatric disorders) | 0 | 1 | 2
Depressed mood (Psychiatric disorders) | 0 | 0 | 1
Hallucination (Psychiatric disorders) | 0 | 0 | 1
Major depression (Psychiatric disorders) | 0 | 0 | 1
Mental status changes (Psychiatric disorders) | 2 | 2 | 4
Mixed anxiety and depressive disorder (Psychiatric disorders) | 1 | 0 | 0
Suicidal ideation (Psychiatric disorders) | 0 | 0 | 2
Acute kidney injury (Renal and urinary disorders) | 16 | 13 | 34
Chronic kidney disease (Renal and urinary disorders) | 0 | 0 | 7
End stage renal disease (Renal and urinary disorders) | 1 | 0 | 3
Glomerulonephritis (Renal and urinary disorders) | 0 | 0 | 1
Haematuria (Renal and urinary disorders) | 3 | 3 | 8
Haemorrhage urinary tract (Renal and urinary disorders) | 0 | 0 | 1
Hydronephrosis (Renal and urinary disorders) | 0 | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 1 | 1 | 1
Nephrotic syndrome (Renal and urinary disorders) | 0 | 0 | 1
Polyuria (Renal and urinary disorders) | 0 | 0 | 1
Renal disorder (Renal and urinary disorders) | 0 | 0 | 1
Renal failure (Renal and urinary disorders) | 1 | 0 | 5
Renal impairment (Renal and urinary disorders) | 0 | 2 | 7
Renal pseudoaneurysm (Renal and urinary disorders) | 0 | 0 | 1
Ureteric obstruction (Renal and urinary disorders) | 1 | 0 | 0
Ureterolithiasis (Renal and urinary disorders) | 0 | 0 | 3
Urinary retention (Renal and urinary disorders) | 3 | 0 | 7
Urinary tract obstruction (Renal and urinary disorders) | 0 | 0 | 1
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1 | 0 | 5
Breast pain (Reproductive system and breast disorders) | 1 | 0 | 0
Prostatitis (Reproductive system and breast disorders) | 0 | 0 | 2
Prostatomegaly (Reproductive system and breast disorders) | 0 | 0 | 1
Scrotal swelling (Reproductive system and breast disorders) | 0 | 0 | 1
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 3 | 1 | 7
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 3
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 | 1 | 13
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 5
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 3
Hypercapnia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 2
Organising pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 3 | 4 | 10
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2
Pulmonary alveolar haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 3
Pulmonary amyloidosis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 4
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 3
Pulmonary infarction (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 7
Pulmonary toxicity (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 12
Actinic keratosis (Skin and subcutaneous tissue disorders) | 2 | 0 | 0
Cellulite (Skin and subcutaneous tissue disorders) | 0 | 0 | 2
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Eczema (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 2
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Rash papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Skin necrosis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Stasis dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Cardiac ablation (Surgical and medical procedures) | 0 | 0 | 1
Implantable defibrillator insertion (Surgical and medical procedures) | 0 | 0 | 1
Muscle electrostimulation therapy (Surgical and medical procedures) | 0 | 0 | 1
Therapy change (Surgical and medical procedures) | 0 | 1 | 0
Wound treatment (Surgical and medical procedures) | 0 | 0 | 1
Aortic dissection (Vascular disorders) | 0 | 0 | 1
Aortic stenosis (Vascular disorders) | 0 | 1 | 10
Arteriovenous fistula (Vascular disorders) | 1 | 0 | 0
Axillary vein thrombosis (Vascular disorders) | 1 | 0 | 0
Bleeding varicose vein (Vascular disorders) | 0 | 1 | 0
Circulatory collapse (Vascular disorders) | 0 | 0 | 2
Distributive shock (Vascular disorders) | 0 | 0 | 1
Embolism (Vascular disorders) | 0 | 0 | 1
Embolism venous (Vascular disorders) | 0 | 0 | 1
Extremity necrosis (Vascular disorders) | 0 | 0 | 1
Haematoma (Vascular disorders) | 2 | 0 | 2
Haemorrhage (Vascular disorders) | 0 | 1 | 0
Hypertensive emergency (Vascular disorders) | 0 | 0 | 1
Hypertensive urgency (Vascular disorders) | 0 | 0 | 1
Hypotension (Vascular disorders) | 2 | 4 | 16
Iliac artery stenosis (Vascular disorders) | 1 | 0 | 0
Ischaemic limb pain (Vascular disorders) | 1 | 0 | 0
Pelvic venous thrombosis (Vascular disorders) | 1 | 0 | 0
Peripheral arterial occlusive disease (Vascular disorders) | 0 | 1 | 2
Peripheral artery occlusion (Vascular disorders) | 0 | 0 | 2
Peripheral artery stenosis (Vascular disorders) | 1 | 0 | 1
Peripheral embolism (Vascular disorders) | 0 | 0 | 3
Peripheral ischaemia (Vascular disorders) | 0 | 0 | 2
Peripheral vein stenosis (Vascular disorders) | 0 | 0 | 1
Peripheral venous disease (Vascular disorders) | 0 | 0 | 1
Shock (Vascular disorders) | 1 | 0 | 1
Shock haemorrhagic (Vascular disorders) | 1 | 0 | 1
Subclavian vein thrombosis (Vascular disorders) | 1 | 0 | 0
Thrombosis (Vascular disorders) | 1 | 0 | 1
Venous thrombosis limb (Vascular disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort A: Tafamidis (Parent and Extension Study) (N=170) | Cohort A: Placebo (Parent Study)/Tafamidis (Extension Study) (N=82) | Cohort B: Tafamidis (Only in Extension Study) (N=1476)
Anaemia (Blood and lymphatic system disorders) | 14 | 12 | 78
Leukocytosis (Blood and lymphatic system disorders) | 1 | 5 | 2
Atrial fibrillation (Cardiac disorders) | 32 | 17 | 150
Cardiac failure (Cardiac disorders) | 22 | 9 | 167
Pericardial effusion (Cardiac disorders) | 6 | 6 | 8
Ventricular tachycardia (Cardiac disorders) | 10 | 9 | 20
Cataract (Eye disorders) | 10 | 1 | 24
Abdominal pain upper (Gastrointestinal disorders) | 5 | 5 | 20
Ascites (Gastrointestinal disorders) | 9 | 4 | 19
Constipation (Gastrointestinal disorders) | 18 | 15 | 117
Diarrhoea (Gastrointestinal disorders) | 15 | 8 | 97
Dysphagia (Gastrointestinal disorders) | 11 | 7 | 29
Nausea (Gastrointestinal disorders) | 17 | 10 | 48
Vomiting (Gastrointestinal disorders) | 10 | 7 | 30
Asthenia (General disorders) | 13 | 12 | 54
Fatigue (General disorders) | 19 | 15 | 78
Gait disturbance (General disorders) | 5 | 6 | 10
Oedema peripheral (General disorders) | 26 | 18 | 100
Peripheral swelling (General disorders) | 9 | 5 | 22
Pyrexia (General disorders) | 6 | 5 | 23
Congestive hepatopathy (Hepatobiliary disorders) | 1 | 5 | 6
Bronchitis (Infections and infestations) | 9 | 6 | 38
Cellulitis (Infections and infestations) | 16 | 8 | 51
Nasopharyngitis (Infections and infestations) | 9 | 6 | 30
Pneumonia (Infections and infestations) | 10 | 12 | 38
Upper respiratory tract infection (Infections and infestations) | 12 | 2 | 53
Urinary tract infection (Infections and infestations) | 18 | 16 | 75
Contusion (Injury, poisoning and procedural complications) | 13 | 5 | 40
Fall (Injury, poisoning and procedural complications) | 41 | 34 | 146
Limb injury (Injury, poisoning and procedural complications) | 7 | 5 | 24
Skin abrasion (Injury, poisoning and procedural complications) | 11 | 6 | 25
Skin laceration (Injury, poisoning and procedural complications) | 12 | 13 | 46
Wound (Injury, poisoning and procedural complications) | 4 | 5 | 13
Blood creatinine increased (Investigations) | 2 | 5 | 14
Gamma-glutamyltransferase increased (Investigations) | 3 | 6 | 13
Weight decreased (Investigations) | 10 | 8 | 32
Decreased appetite (Metabolism and nutrition disorders) | 9 | 8 | 50
Dehydration (Metabolism and nutrition disorders) | 9 | 4 | 21
Fluid retention (Metabolism and nutrition disorders) | 9 | 3 | 19
Gout (Metabolism and nutrition disorders) | 18 | 10 | 113
Hyperglycaemia (Metabolism and nutrition disorders) | 2 | 6 | 10
Hyperkalaemia (Metabolism and nutrition disorders) | 5 | 5 | 35
Hyperuricaemia (Metabolism and nutrition disorders) | 9 | 5 | 32
Hypervolaemia (Metabolism and nutrition disorders) | 10 | 11 | 76
Hypokalaemia (Metabolism and nutrition disorders) | 23 | 17 | 61
Hyponatraemia (Metabolism and nutrition disorders) | 11 | 13 | 35
Arthralgia (Musculoskeletal and connective tissue disorders) | 29 | 12 | 78
Back pain (Musculoskeletal and connective tissue disorders) | 18 | 12 | 65
Muscle spasms (Musculoskeletal and connective tissue disorders) | 14 | 4 | 53
Muscular weakness (Musculoskeletal and connective tissue disorders) | 11 | 7 | 19
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 12 | 9 | 20
Pain in extremity (Musculoskeletal and connective tissue disorders) | 24 | 9 | 55
Balance disorder (Nervous system disorders) | 11 | 4 | 16
Dizziness (Nervous system disorders) | 24 | 11 | 97
Anxiety (Psychiatric disorders) | 7 | 6 | 28
Depression (Psychiatric disorders) | 8 | 8 | 23
Insomnia (Psychiatric disorders) | 13 | 13 | 57
Acute kidney injury (Renal and urinary disorders) | 15 | 15 | 54
Chronic kidney disease (Renal and urinary disorders) | 10 | 13 | 20
Haematuria (Renal and urinary disorders) | 7 | 11 | 47
Renal failure (Renal and urinary disorders) | 11 | 3 | 10
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 3 | 5 | 21
Cough (Respiratory, thoracic and mediastinal disorders) | 29 | 18 | 81
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 31 | 18 | 110
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 13 | 5 | 38
Orthopnoea (Respiratory, thoracic and mediastinal disorders) | 6 | 5 | 11
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 23 | 24 | 58
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 2 | 5 | 8
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 3 | 7 | 9
Pruritus (Skin and subcutaneous tissue disorders) | 17 | 8 | 36
Skin ulcer (Skin and subcutaneous tissue disorders) | 10 | 3 | 25
Hypotension (Vascular disorders) | 14 | 20 | 70

LIMITATIONS AND CAVEATS:
For analyses in current extension study for Cohort A based on CMA set, it combined data from participants in parent study B3461028, including participants who died, discontinued in parent study B3461028, or did not enroll into the current extension study B3461045.Data for these participants is used only in few planned outcomes and these participants do not reflect in any other section of this record. For reference, results for B3461028 can be found at ClinicalTrails.gov with NCT ID: NCT01994889.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publication until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2020-01-24): https://cdn.clinicaltrials.gov/large-docs/30/NCT02791230/Prot_000.pdf
  • Statistical Analysis Plan (2021-03-11): https://cdn.clinicaltrials.gov/large-docs/30/NCT02791230/SAP_001.pdf